CLINICAL TRIAL: NCT06365632
Title: A Prospective, Randomized, Parallel, Single-blind Clinical Study of the Effectiveness, Tolerability and Safety of the Drug "Anti-spike, Gel, 100 g in Bottles in Package No. 1" Produced by the Republican Unitary Enterprise "Unitekhprom BSU", Belarus, With a Single Intraperitoneal Use After Surgical Interventions in Adult Patients With Acute Phlegmonous Appendicitis
Brief Title: Clinical Study of the Effectiveness, Tolerability and Safety of the Drug "Anti-spike, Gel, 100 g in Bottles in Package No. 1" Produced by the Republican Unitary Enterprise "Unitekhprom BSU", With a Single Intraperitoneal Use After Surgery in Adult Patients With Acute Phlegmonous Appendicitis
Acronym: OLTOSPAN-02
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Research Institute for Physical Chemical Problems of the Belarusian State University (Other)
Collaborators: Unitary Enterprise UNITEHPROM BSU (Unknown); City Clinical Hospital of Emergency Medical Care of Minsk (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: OLTOSPAN-02
Record Dates: First submitted 2024-04-09; First posted 2024-04-15 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Abdominal Adhesions
Keywords: phlegmonous appendicitis; ketorolac tromethamine; gel; abdominal adhesions

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Surgical intervention due to acute phlegmanous appendicitis using the drug antispike (Experimental): Placebo-controlled, single-blind clinical trial of the effectiveness, tolerability and safety of the drug "Antispike, gel, 100 g in a bottle" produced by Unitary Enterprise Unitehprom BGU, Republic of Belarus, in adult patients after surgery for acute phlegmonous appendicitis. An antegrade appendectomy is performed, after which the drug Antispike is used.
  Interventions: Drug: Antispike gel, 100 g in a flask, produced by UNITEHPROM BSU, Republic of Belarus; Procedure: antegrade appendectomy
- surgical intervention due to acute phlegmanous appendicitis (Sham Comparator): An antegrade appendectomy is performed without using Antispike.
  Interventions: Procedure: antegrade appendectomy

INTERVENTIONS:
Drug: Antispike gel, 100 g in a flask, produced by UNITEHPROM BSU, Republic of Belarus — An antegrade appendectomy is performed, after which 50 to 100 ml of Antispike is applied in a thin layer to the surface of the cecum, the surface of adjacent organs and the parietal peritoneum of the right iliac region. The wound is sutured tightly.
  Arms: Surgical intervention due to acute phlegmanous appendicitis using the drug antispike
Procedure: antegrade appendectomy — An antegrade appendectomy is performed without using Antispike.

SUMMARY:
The purpose of the clinical trials is the evaluation of the effectiveness and safety of a single intraperitoneal use of the drug "Antispike, gel, 100 g in a bottle" produced by Unitary Enterprise Unitehprom BSU, Belarus in patients after surgical control of acute phlegmonous appendicitis to prevent abdominal adhesions.

DETAILED DESCRIPTION:
The prospective, randomized, placebo-controlled, single-blind clinical trial of the effectiveness, tolerability and safety of the drug "Antispike, gel, 100 g in a bottle" produced by Unitary Enterprise Unitehprom BGU, Republic of Belarus, in adult patients after surgery for acute phlegmonous appendicitis.

Research objectives:

* To evaluate the immediate, rapid and long-term results of using Antispike as a drug for preventive adhesions in patients who have a medium and high risk factor for the development of adhesions and are undergoing surgery for acute phlegmonous appendicitis;
* Identify the possibility of undesirable effects that may occur when using the drug;
* to conduct a comparative assessment of the immediate results of using the drug Antispike as a means of preventing adhesions in patients with minor phlegmonous appendicitis with an effect in the control group, in patients in whom anti-adhesion drugs were not used;
* Detailed description of the conditions and method of use of the Antispike drug.

ELIGIBILITY:
Inclusion Criteria:

* Presence of acute phlegmonous appendicitis requiring surgical intervention.
* Presence of medium or high risk factor for the development of adhesions of the abdominal cavity;
* Age of patients from 18 to 65 years.
* Absence of severe concomitant diseases in decompensation stage, oncologic diseases, as well as diseases requiring steroid therapy.
* Presence of written informed consent of the patient to participate in the study.
* The patient's ability to fulfill the instructions of the research physician and comply with the study design.

Exclusion Criteria:

* At the subject own request without explaining the reasons for the behavior.
* At the request of the physician-researcher if the subject violates the requirements of the protocol in terms of diet, smoking, consumption of alcoholic beverages, and use of medications without the prescription of the physician-researcher.
* For reasons independent of the subject and the research physician, if the subject has drug intolerance or other life-threatening or life-threatening adverse reactions to drug administration that require emergency pharmacotherapy.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2025-03-19 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Number of patients with acute phlegmonous appendicitis cured | from surgery to 3 weeks
  Number of patients cured

SECONDARY OUTCOMES:
absence of signs of adhesions | from surgery to 4 weeks
  absence of signs of adhesions according to clinical and ultrasound studies

OTHER OUTCOMES:
increase in the sliding distance of the cecum | from surgery to 7 days
  increase in the sliding distance of the cecum, determined by the results of an ultrasound examination on the 7th day after appendectomy

CONTACTS AND LOCATIONS:
Locations (1):
- CITY CLINICAL EMERGENCY HOSPITAL of Minsk, Minsk, Belarus

IPD SHARING:
Plan to Share IPD: Undecided